CLINICAL TRIAL: NCT00706758
Title: Structured Patient Education Versus Written Information for Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Magnus Simrén, Sahlgrenska University Hospital, Gothenburg, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S487-02
Record Dates: First submitted 2008-06-25; First posted 2008-06-30 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2008-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Patient education
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Structured patients group intervention - IBS school
  Interventions: Behavioral: IBS school
- 2 (Active Comparator): Written information - IBS-guidebook
  Interventions: Behavioral: IBS-guidebook

INTERVENTIONS:
Behavioral: IBS school — Structured patient group education
  Arms: 1
Behavioral: IBS-guidebook — Written information - IBS-guidebook
  Arms: 2

SUMMARY:
In this randomized controlled study in patients with irritable bowel syndrome (IBS) we plan to compare the effects of a structured patient group education (IBS school) with receiving only written information in the form of a IBS-guidebook. The effects of the interventions on GI and psychological symptom severity, knowledge and quality of life will be assessed with validated questionnaires at baseline and 3 and 6 months after the intervention.

DETAILED DESCRIPTION:
In this randomized controlled study in patients with irritable bowel syndrome (IBS) we plan to compare the effects of a structured patient group education (IBS school) with receiving only written information in the form of a IBS-guidebook. We plan to include men and women 18 to 70 years old, with IBS according to the Rome II criteria, who are referred from physicians in primary care and secondary/tertiary care to participate in the study. The education will be held at the GI out patient clinic at Sahlgrenska University hospital in Gothenburg. A nurse, specialized in GI functional disorders will conduct an interview with each patient for about 30 minutes to collect additional information from the patients before inclusion. The patients will be informed about the positive results obtained in previous studies with both interventions, i.e. a structured patient education (IBS school) and a self-help guidebook. Patients with an organic GI disease and/or with another disease potentially affecting the GI symptoms were excluded. Likewise, patients with a severe psychiatric disease were excluded due to potential problems to participate in a group intervention. In order to allocate an equal number of patients to both of the interventions during the study, a number of up to 20 patients will be interviewed in a block during one week. After all these interviews the patients will be randomly divided into two groups with an equal number of patients in each group. The groups will then be randomized 1:1 to either start the IBS school within two to three weeks, or to receive the IBS Guidebook. The patients in the guidebook group will be offered to participate in the IBS school six months later, as part of the clinical routine at our unit (as requested by the ethics committee). The effects of the interventions on GI and psychological symptom severity, knowledge and quality of life will be assessed with validated questionnaires at baseline and 3 and 6 months after the intervention:

1. Perceived knowledge about IBS
2. IBS Severity Scoring System (IBS-SSS)
3. IBS Quality of Life (IBSQOL)
4. Visceral Sensitivity Index (VSI)
5. The Hospital Anxiety and Depression Scale (HAD)

The interventions:

IBS school The IBS school is designed based on the self-efficacy theory , and the general theory of nursing. Moreover, the education is performed based on a biopsychosocial model considered to be important in functional GI disorders. The IBS-school consists of six sessions held once per week in a group setting with eight to ten patients in each group. Five different health care professionals (nurse, gastroenterologist, dietician, physiotherapist and psychologist) are involved in the education, in order to cover a wide spectra of issues related to IBS. Each of the professionals will hold one session for two hours where a lot of space is given for discussion in the group. This intervention has been described in detail previously (Ringström et. al. Submitted).

IBS Guidebook The IBS Guidebook consists of two booklets, written for IBS patients by one of the gastroenterologists in this study (MS). The booklets are detailed and cover the same areas of issues related to IBS as are covered in the structured education, namely pathophysiological mechanisms, GI and extra intestinal symptoms, the diagnostic workup, treatment options, food related issues, psychological and lifestyle factors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 70 years old, with IBS according to the Rome II criteria
* Written informed consent

Exclusion Criteria:

* An organic GI disease and/or with another disease potentially affecting the GI symptoms
* Severe psychiatric disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2004-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Effect on GI symptoms as measured by IBS-SSS | Basleline and 3 and 6 months

SECONDARY OUTCOMES:
Effects on Quality of life (IBSQOL), Psychological symptoms (HAD), GI specific anxiety (VSI) and knowledge about IBS. | Baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden